CLINICAL TRIAL: NCT00365300
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Treatment-Withdrawal Study of the Efficacy and Safety of Pantoprazole Sodium Enteric-Coated Granules in Infants (1 Through 11 Months) With Symptomatic GERD.
Brief Title: Study Evaluating the Efficacy and Safety of Pantoprazole in Infants With Symptomatic Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3001B3-329
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Results first posted 2010-01-07 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-04

CONDITIONS: Gastroesophageal Reflux
Keywords: GERD; Infants; Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Pantoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Pantoprazole (Active Comparator)
  Interventions: Drug: pantoprazole
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pantoprazole
  Arms: Pantoprazole
Drug: Placebo
  Arms: Placebo

SUMMARY:
To assess the efficacy of pantoprazole for the treatment of infants with symptomatic Gastroesophageal Reflux Disease (GERD).

ELIGIBILITY:
Inclusion Criteria:

* term or post term infants beyond the neonatal period of an age greater than 28 days but less than or equal to 11 months
* clinical diagnosis of GERD
* weight greater than 2.5 kg and less than or equal to 15 kg

Exclusion Criteria:

* known history of upper GI anatomic disorders
* history of acute life-threatening medical conditions
* clinically significant medical conditions or laboratory abnormalities

Ages: 28 Days to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2006-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (38):
- United States (38):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Oakland, California
  - Orange, California
  - Washington D.C., District of Columbia
  - Miami, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Peoria, Illinois
  - Bardstown, Kentucky
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Flint, Michigan
  - Jackson, Mississippi
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Camden, New Jersey
  - Mays Landing, New Jersey
  - Morristown, New Jersey
  - Brooklyn, New York
  - Buffalo, New York
  - Valhalla, New York
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Bethlehem, Pennsylvania
  - Memphis, Tennessee
  - Temple, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Norfolk, Virginia
  - Richmond, Virginia
  - Huntington, West Virginia
  - Morgantown, West Virginia
  - Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited worldwide from September 2006 to August 2007.
Pre-assignment Details: Patients were screened for 2 weeks and provided non-pharmacologic conservative therapy including hypoallergenic formula thickened with rice cereal. Patients who improved on this treatment were not eligible for enrollment.
Groups:
- Pantoprazole Sodium Granules: Double Blind Treatment-withdrawal phase (weeks 5-8) Pantoprazole sodium granules at a dose of approximately 1.2 mg/kg daily (5 mg for weight < 7 kg or 10 mg for weight ≥ 7 kg) in an oral suspension. An Open Label Treatment run-in phase (weeks 1-4) preceded the Double Blind Treatment-withdrawal phase and patients received: Pantoprazole sodium granules at a dose of approximately 1.2 mg/kg daily (5 mg for weight < 7 kg or 10 mg for weight ≥7 kg) in an oral suspension.
- Placebo: Double Blind Treatment-withdrawal phase (weeks 5-8): Matching placebo. An Open Label Treatment run-in phase (weeks 1-4) preceded the Double Blind Treatment-withdrawal phase and patients received Pantoprazole sodium granules at a dose of approximately 1.2 mg/kg daily (5 mg for weight < 7 kg or 10 mg for weight ≥7 kg) in an oral suspension.
Period: Open-label Phase
Arm/Group | Pantoprazole Sodium Granules | Placebo
Started | 129 | 0
Completed | 107 | 0
Not Completed | 22 | 0
Not completed — Adverse Event | 4 | 0
Not completed — Failed to Return | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Noncompliance | 9 | 0
Not completed — Parent/Legal Guardian Request | 4 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Patient skipped open label phase | 1 | 0
Period: Double-blind Phase
Arm/Group | Pantoprazole Sodium Granules | Placebo
Started | 54 | 54
Completed | 43 | 45
Not Completed | 11 | 9
Not completed — Failed to return | 1 | 0
Not completed — Noncompliance | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 3 | 1
Not completed — Lack of Efficacy | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pantoprazole Sodium Granules | Placebo | Total
Number analyzed (Participants) | 52 | 54 | 106
Age Continuous [Mean (Standard Deviation); unit: months] | 5.15 (2.81) | 5.04 (2.81) | 5.09 (2.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 34 | 34 | 68

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Withdrawn From Study Due to Lack of Efficacy.
Description: Lack of efficacy defined as 1 or more of the following occurring during the double blind treatment-withdrawal phase: significant worsening of gastroesophageal reflux disease (GERD) symptoms frequency, a diagnostic test (e.g., endoscopy) demonstrating worsening of esophagitis, maximal antacid intake for ≥ 7 continuous days, or severe GERD symptoms based on physician's judgment.
Time Frame: 4 weeks double-blind
Population: The analysis population was the Modified Intent to Treat, which included all GERD patients who completed the 4 week open-label treatment phase, were randomized into the 4 week double-blind phase, and took at least one dose of double-blind treatment.
Measure: Number; unit: patients
Arm/Group | Pantoprazole Sodium Granules | Placebo
Number analyzed (Participants) | 52 | 54
patients | 6 | 6
Statistical Analysis 1: Comparison: Pantoprazole Sodium Granules vs Placebo; Test type: Superiority or Other; p = 1.0, Fisher Exact; Risk Difference (RD) = 0.004

ADVERSE EVENTS:
Arm/Group | Screening | Pantoprazole Sodium Granules (Open-Label Phase) | Pantoprazole Sodium Granules (Double-blind Phase) | Placebo (Double-blind Phase) | Follow-up
Serious Adverse Events (participants affected / at risk) | 2/129 | 4/128 | 0/54 | 1/54 | 3/127
Other Adverse Events (participants affected / at risk) | 52/129 | 85/128 | 28/54 | 28/54 | 25/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Screening (N=129) | Pantoprazole Sodium Granules (Open-Label Phase) (N=128) | Pantoprazole Sodium Granules (Double-blind Phase) (N=54) | Placebo (Double-blind Phase) (N=54) | Follow-up (N=127)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Otitis media (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Screening (N=129) | Pantoprazole Sodium Granules (Open-Label Phase) (N=128) | Pantoprazole Sodium Granules (Double-blind Phase) (N=54) | Placebo (Double-blind Phase) (N=54) | Follow-up (N=127)
Accidental injury (General disorders) | 1 | 1 | 1 | 2 | 1
Fever (General disorders) | 10 | 15 | 3 | 2 | 0
Flu syndrome (General disorders) | 0 | 1 | 1 | 0 | 0
Infection (General disorders) | 3 | 4 | 0 | 1 | 0
Lab test abnormal (General disorders) | 0 | 1 | 0 | 1 | 0
Moniliasis (General disorders) | 1 | 0 | 0 | 1 | 0
Anorexia (Gastrointestinal disorders) | 0 | 3 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 5 | 1 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 14 | 2 | 2 | 1
Oral moniliasis (Gastrointestinal disorders) | 2 | 7 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 7 | 3 | 2 | 3
Creatine phosphokinase increased (Metabolism and nutrition disorders) | 1 | 1 | 3 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hyperlipidemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Anxiety (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Emotional lability (Nervous system disorders) | 0 | 2 | 1 | 0 | 0
Sleep disorder (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Twitching (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 0
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 1 | 2
Cough increased (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 2 | 4 | 1
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0/128 | 2 | 1 | 0 | 2
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 12 | 3 | 1 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 14 | 29 | 9 | 8 | 6
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Contact dermatitis (Skin and subcutaneous tissue disorders) | 5 | 8 | 2 | 0 | 0
Cutaneous moniliasis (Skin and subcutaneous tissue disorders) | 1 | 5 | 1 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 5 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 0
Furunculosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Impetigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 4 | 3 | 2 | 1
Seborrhea (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 2 | 0 | 1 | 1
Otitis media (Ear and labyrinth disorders) | 2 | 13 | 3 | 0 | 4
Urinary tract infection (Renal and urinary disorders) | 4 | 0 | 0 | 2 | 2
Tooth disorder (Gastrointestinal disorders) | 0 | 5 | 0 | 2 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 4 | 0 | 0 | 0
Hematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Abdominal pain (General disorders) | 0 | 1 | 0 | 0 | 0
Hernia (General disorders) | 0 | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
SGOT increased (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
SGPT increased (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Agitation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Nervousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Fungal dermatitis (Skin and subcutaneous tissue disorders) | 0 | 5 | 0 | 0 | 0
Maculopapular rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Testis disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Vulvovaginal disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.